CLINICAL TRIAL: NCT02983747
Title: Autologous Platelet Rich Plasma in Ultrasound Guided Intervertebral Disk Injection Therapy for Chronic Low Back Pain
Brief Title: Autologous Platelet Rich Plasma on Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Xuhua Lu, Vice Director of Spine Surgery, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201540379
Record Dates: First submitted 2016-11-21; First posted 2016-12-06 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Low Back Pain
Keywords: Platelet Rich Plasma; Intervertebral Disk Injection Therapy; Low Back Pain; Ultrasound Guided; Degenerative Spinal Disease
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP Treatment(P) (Experimental): PRP intra-disk injection therapy combined with NSAIDs medication (Loxoprofen Sodium tablets).
  Interventions: Other: PRP Treatment(P); Drug: Medication Treatment(Loxoprofen Sodium tablets,M)
- Medication Treatment(M) (Active Comparator): NSAIDs medication(Loxoprofen Sodium tablets) therapy only.
  Interventions: Drug: Medication Treatment(Loxoprofen Sodium tablets,M)

INTERVENTIONS:
Other: PRP Treatment(P) — Ultrasound(Philips® iU22 ultrasound system) guided intra-disk injection using 2 ml of platelet rich plasma, containing 0.2 ml of calcium chloride(SINE®, SHANGHAI XINYI PHARMACEUTIAL Co . Ltd .) per treatment
  Other Names: Platelet Rich Plasma
  Arms: PRP Treatment(P)
Drug: Medication Treatment(Loxoprofen Sodium tablets,M) — Loxoprofen Sodium tablets(LOXONNIN®, DAICHI SANKYO PHARMACEUTIAL (SHANGHAI) Co . Ltd .)，P.O., 60mg, three times a day
  Other Names: LOXONNIN®, DAICHI SANKYO PHARMACEUTIAL (SHANGHAI) Co . Ltd .

SUMMARY:
The purpose of this study is to evaluate the effectiveness of autologous platelet-rich plasma (PRP) injection therapy for low back pain patients. Our hypothesis is that PRP will reduce the pain feeling and benefit for restore of the intervertebral disk.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain more than 2months
* Visual analog scale score more than 4
* Positive X-ray, MRI or CT scan findings
* Pfirrmann grading I-III
* Well understanding and communication ability

Exclusion Criteria:

* History of allergy
* Hemorrhagic trend or use of anticoagulant therapy
* Mental diseases
* Active infection or recent infectious diseases within 3 months
* Local skin infection near the puncture location
* Severe lumbar spinal stenosis, lumbar spondylolisthesis, ossification of posterior longitudinal
* Ligament and lumbar disc herniation（more than 5mm）
* Immunologic diseases
* Tumors
* Metastatic disease
* Recent surgery less than 3 months)
* Pregnancy

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) | 1 year
  Pain relief evaluated using change from baseline in Visual Analog Scale (VAS):baseline, 1 week ,and 1 month, 2 months, 6 months, 12 months after intervention.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | 1 year
  Pain relief and functions evaluated using change from baseline in Oswestry Disability Index (ODI): baseline, 1 week ,and 1 month, 2 months, 6 months, 12 months after intervention.
Functional Rating Index | 1 year
  Spinal functions evaluated using change from baseline by Functional Rating Index: baseline, 1 week ,and 1 month, 2 months, 6 months, 12 months after intervention.
Measuring the Quality of life using SF-36 questionnaire | 1 year
  Functions evaluated using change from baseline in SF-36:baseline, 1 week ,and 1 month, 2 months, 6 months, 12 months after intervention.
Imaging change | 1 year
  Imaging change by MRI scan: : baseline, 1 month, 6 months, 12 months after intervention.
Number of patients with side effect | Within 1 year after injection therapy
  Record how many patients had side effects after intervention (eg.aggravation of pain*(VAS change increased more than 3 from baseline),anaphylaxis,sensory/motion disturbances).

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Lu, M.D., Principal Investigator — Shanghai Changzheng Hospotal
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided